CLINICAL TRIAL: NCT02628119
Title: Access Flow Based Intervention for Management of Arteriovenous Hemodialysis Access Dysfunction. A Prospective Randomized Controlled Study.
Brief Title: Access Flow Based Intervention for Management of Arteriovenous Hemodialysis Access Dysfunction.
Acronym: FBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Naveed Ul Haq, Director Interventional Nephrology and Dialysis Access Program, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2151 040
Record Dates: First submitted 2015-11-19; First posted 2015-12-11 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Hemodialysis Arteriovenous Fistula Maturation Failure
Keywords: Hemodialysis; vascular access; access flow

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-procedural access flow (Experimental): Management of access dysfunction based on intra-procedure access flow monitoring.
  Criteria for target access flow:
  Within 90% of baseline access flow if known 180% increase from pre-intervention flow if access flow not known 600ml/min for thrombosed grafts and 500 ml/min for thrombosed arteriovenous fistula in case baseline access flow not known
  Interventions: Procedure: Intra-procedural access flow
- Standard Angioplasty (Active Comparator): Intervention based on current standards of care i.e. 2 dimensional angiographic views.
  Interventions: Procedure: Standard Angioplasty

INTERVENTIONS:
Procedure: Intra-procedural access flow — Intra-procedure access flow technique:
  Room temperature saline is injected into the vascular access blood stream during angioplasty via ReoCath(tm) 6 French antegrade or retrograde flow catheters. When the saline is injected into the access, an injection thermistor located close to the proximal end of the catheter records the temperature of the injected saline. A second thermistor located close to the distal tip of the catheter then records the thermodilution within the access and the HVT100 endovascular flow meter calculates and displays intragraft blood flow in ml/min.
  Arms: Intra-procedural access flow
Procedure: Standard Angioplasty — Intervention based on 2 Dimensional fluoroscopy views
  Arms: Standard Angioplasty

SUMMARY:
Hemodialysis (HD) vascular access dysfunction is a huge clinical problem which results in significant clinical morbidity in patients with End Stage Renal Disease (ESRD), causing a severe economic burden on any health care system. Arteriovenous (A-V) dialysis accesses are the preferred form of permanent dialysis access as compared to central venous catheters (CVC) . One of the reasons for CVC use is poor long term patency rates of A-V access. Arteriovenous Grafts (AVG) have a primary patency rates of just under 50% at 12 months and around 33% at 18 months. Native arteriovenous fistula (AVF) are slightly better with primary patency rates of around 60 percent at one year and 51 percent at 2 years. The most common cause for AVF and AVG dysfunction is stenosis development due to neointimal hyperplasia (NIH) within the circuit leading to access thrombosis. Percutaneous transluminal angioplasty (PTA) is the current standard of treatment for these lesions. Despite being the treatment of choice for these lesions patency rates after PTA continue to be dismal. One of the problems with poor long term outcomes after successful intervention is how you assess immediate intervention success. Successful angioplasty is defined by Dialysis Outcome Quality Initiative (DOQI) guidelines as one where only less than 30% residual stenosis remains at the end of intervention. Unfortunately angiographic images post angioplasty correlate poorly with improvement of access flows through the arteriovenous circuit. There are two main problems with these practice standards. First, they are based on a 2-dimensional angiographic view of the lesion which may be misleading. Secondly, this assessment of recoil is very subjective and not base on objective data.

Access flow monitoring can now be performed intra-procedurally with thermal dilution technique. Its benefit was shown in a small pilot study. To date there have not been any randomized controlled trials to assess the benefit of such an approach where intervention is based on improvements in access flow at the time of intervention. We hypothesize that such an approach will improve outcomes after interventions related to access dysfunction. This may also identify the right scenarios in which stent placement may benefit thus improving outcomes after stent placement as well.

DETAILED DESCRIPTION:
Background:

The number of patients with End Stage Renal Disease (ESRD) requiring renal replacement therapy (RRT) in the form of dialysis is on the rise. Hemodialysis (HD) remains the most prevalent form of RRT for patients with ESRD. Just in the United States there are more than 350,000 patients with ESRD on hemodialysis (HD) and the number is expected to increase to 500,000 by the year 2023. Recent data provided by Saudi Centre for Organ Transplantation shows that there are just over 13000 patients with ESRD on hemodialysis in the Kingdom of Saudi Arabia (KSA). This number is expected to rise at a rate of 7-8% annually reaching 18000 by year 2018. Establishing a viable vascular access is crucial and is considered the 'life-line' for such patients.

HD vascular access dysfunction is a huge clinical problem which results in significant clinical morbidity in patients with ESRD, causing a severe economic burden on any health care system. In the United States <50% of all hemodialysis accesses remain patent at 3 years with the economic burden of maintaining vascular access patency calculated to exceed $1 billion annually. Arteriovenous (A-V) dialysis accesses are the preferred form of permanent dialysis access as compared to central venous catheters (CVC) due to less complications and better patient outcomes. Native arteriovenous fistulae (AVF) and synthetic arteriovenous grafts (AVG) are the two main types of A-V access used for HD. Despite the obvious benefits many patients on HD continue to dialyze with CVC as there dialysis access. One of the reasons for CVC use is poor long term patency rates of A-V access. AVG have a primary patency rates of just under 50% at 12 months and around 33% at 18 months. AVF are slightly better with primary patency rates of around 60 percent at one year and 51 percent at 2 years. The most common cause for AVF and AVG dysfunction is stenosis development due to neointimal hyperplasia (NIH) within the circuit leading to access thrombosis. Percutaneous transluminal angioplasty (PTA) is the current standard of treatment for these lesions. Despite being the treatment of choice for these lesions patency rates after PTA continue to be dismal. Long-term success rates are generally listed as either primary/unassisted rates (patency without additional procedures)) or secondary/assisted patency (patency with additional procedures). Unassisted patency rates for angioplasty generally range from 41 to 76 percent at six months and 31 to 45 percent at one year. To improve the primary patency after intervention many strategies have been looked at. Placement of covered stents at the time of intervention has been used, but patency rates after stent placements although better than PTA, are still not optimal. One of the problems with poor long term outcomes after successful intervention is how you assess immediate intervention success. Successful angioplasty is defined by Dialysis Outcome Quality Initiative (DOQI) guidelines as one where less than 30% residual stenosis remains at the end of intervention. It is suggested that if residual stenosis is >30% after angioplasty with adequately sized fully effaced angioplasty balloon than stent placement should be considered. Unfortunately angiographic images post angioplasty correlate poorly with improvement of access flows through the arteriovenous circuit. There are two main problems with these practice standards. First, this is based on a 2-dimensional angiographic view of the lesion which may be misleading. Secondly, this assessment of recoil is very subjective and not base on objective data.

Surveillance of AV access with access flow monitoring is recommended to identify AV access with stenosis before they develop thrombosis. One of the methods most commonly used to assess access flows is ultrasound dilution technique. This can be performed at the time of dialysis by trained staff to assess access flows. Access flow measurements are usually done monthly in units who have access surveillance programs in place. It has been shown that improvement in access flows after intervention from baseline or pre intervention values can predict long term outcomes after intervention. Although helpful, but access flows are performed at HD unit on the following days after the patient had intervention. At that time it is impractical to bring the patient back for intervention and leads to additional cost and inconvenience. As such the clinical benefit of this approach is minimal. In addition many dialysis units do not have access flow measurement available and no surveillance programs implemented. Unfortunately this is true for most hemodialysis units in the Kingdom of Saudi Arabia (KSA). Fortunately access flow monitoring can now be performed intra-procedurally with the same ultrasound dilution technique. Its benefit was shown in a small pilot study. To date there have not been any randomized controlled trials to assess the benefit of such an approach where intervention is based on improvements in access flow at the time of intervention. The researchers hypothesize that such an approach will improve outcomes after interventions related to access dysfunction. This may also identify the right scenarios in which stent placement may benefit thus improving outcomes after stent placement as well. This approach should also improve outcomes and reduce repeat hospital visits in areas where access flow monitoring at HD units is not readily available as is the case in most centers in the Kingdom of Saudi Arabia.

Specific Aims In a randomized, controlled, blinded trial the researchers would like to assess the clinical utility of an access flow based intervention approach as compared to conventional approach for managing dialysis arteriovenous access dysfunction.

Materials and Methods

A. Study Design:

Prospective, Randomized Controlled, single centre trial comparing access flow based intervention versus conventional standard approach for dialysis access dysfunction.

B. Study Subjects ESRD patients on HD referred for access dysfunction to the interventional nephrology service at King Faisal Specialist Hospital and Research Center in Riyadh, KSA.

Sample Size:

116 patients are required to have an 80% chance of detecting, at significance level of 5%, an increase in the primary patency outcome measure from 45% in the control group to 70% in the experimental group at 6 months meaning 58 patients in each arm. The researchers plan to enroll a total of 140 patients with 70 in each group.

Data Collection:

Patient Demographics:

Age Sex ESRD or Chronic Kidney Disease stage 5 needing HD Currently on Dialysis Y N

If yes: currently used access type:

Years on Dialysis:

Diabetes Mellitus Hypertension Peripheral Vascular Disease Smoking Coronary artery disease Cerebrovascular accidents Antiplatelet medications

Location of AVF:

Location of AVG:

Reason for procedure: Excessive bleeding post HD Low Access flows High venous or low arterial pressures Physical Examination abnormality Other

Pre-procedure within 3 month baseline access flows known Y N

If known, Value:

Data on 1st Angiogram:

Stenosis present: Y N If yes: Location of Stenosis: Arterial Juxta anastomosis Arterial 1/3rd Middle 1/3rd Venous 1/3rd or venous outflow

Pre-intervention access flow in case of no thrombosis (A):

Targeted access flow:

Stenosis successfully treated radiologically Y N Targeted access flow successfully reached: Y N

Post-intervention access flow (B):

Percentage access flow reached of target (B/A x 100):

Residual Stenosis in %:

By Operator By Blinded Interpreter:

Max diameter of balloon used:

Max inflation pressure of balloon used:

Stent used: Y N

If used, size of stent: # of stent:

Follow up:

Access Flows:

Within 1st three treatments post intervention 3rd month 6th month

Physical Examination abnormalities if any:

3rd month 6th month

Time to first intervention after initial procedure:

If intervention, reason for the need of intervention:

Primary patency at 6 months: Y N

If no, exact duration of primary patency:

Secondary patency at 6 months: Y N

Statistical Considerations:

The researchers will use block-randomization for the recruited subjects into the two arms. Researchers will take the risk difference as an effect measure. The chi-square test will be used to assess the superiority of the new treatment as compared to the standard protocol. Researchers will set the type I error rate at 5%. Baseline comparisons between the two groups will be conducted using the two independent samples t-test for continuous data which will be summarized as means ± standard deviation, and using the chi-square test for categorical data.

Ethical Considerations / Consent Documents The proposal of this study has been approved by the local review authority which is the Office of Research Affairs at King Faisal Specialist Hospital and Research Centre.

All participants will be assigned serial numbers in order of data collection. Each medical record number will be assigned a specific serial number and this list will be kept in the PI's office. All investigators mentioned in the study will have access to them. Databases created will be password protected.

The study will be managed by the PI in cooperation with other Co-Investigators

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with ESRD and access dysfunction secondary to stenosis anywhere in the AVF.

Exclusion Criteria:

* Patients on anti-coagulation and those with bleeding disorders
* Life expectancy less than 12 months.
* Documented severe contrast allergy.
* Inability to come for timely and adequate follow up.
* Patients undergoing transplantation work up and expected to be transplanted within 6 months.
* AVG with access dysfunction developing within 30 days of surgery.
* AVF with early fistula failure.
* Recurrence of stenosis within 3 months of previous intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Primary un-assisted patency | 6 months
  The AVF is still being used for dialysis with a minimum blood pump speed of 300ml/min and no additional procedures have been done to maintain patency

SECONDARY OUTCOMES:
Secondary or assisted patency | 6 months
  The AVF is still being used for dialysis with a minimum blood pump speed of 300ml/min and additional procedures have been done to maintain patency
Number of procedures required in each group to maintain patency | 6 months
  endovascular procedures like angioplasty, stenting, or thrombectomy

CONTACTS AND LOCATIONS:
Overall Officials: Naveed U Haq, MD, FASN, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Foley RN, Collins AJ. The USRDS: what you need to know about what it can and can't tell us about ESRD. Clin J Am Soc Nephrol. 2013 May;8(5):845-51. doi: 10.2215/CJN.06840712. Epub 2012 Nov 2. PMID 23124788
- [Background] Feldman HI, Kobrin S, Wasserstein A. Hemodialysis vascular access morbidity. J Am Soc Nephrol. 1996 Apr;7(4):523-35. doi: 10.1681/ASN.V74523. PMID 8724885
- [Background] Beathard GA. Percutaneous transvenous angioplasty in the treatment of vascular access stenosis. Kidney Int. 1992 Dec;42(6):1390-7. doi: 10.1038/ki.1992.431. PMID 1474770
- [Background] Glanz S, Gordon DH, Butt KM, Hong J, Lipkowitz GS. The role of percutaneous angioplasty in the management of chronic hemodialysis fistulas. Ann Surg. 1987 Dec;206(6):777-81. doi: 10.1097/00000658-198712000-00015. PMID 2961315
- [Background] Ahya SN, Windus DW, Vesely TM. Flow in hemodialysis grafts after angioplasty: Do radiologic criteria predict success? Kidney Int. 2001 May;59(5):1974-8. doi: 10.1046/j.1523-1755.2001.0590051974.x. PMID 11318971
- [Background] Maursetter L, Yevzlin AS. The use of intravascular ultrasound to assist angiography in diagnosis and management of hemodialysis access. Semin Dial. 2011 Jan-Feb;24(1):89-91. doi: 10.1111/j.1525-139X.2011.00840.x. PMID 21338398
- [Background] Krivitski NM, MacGibbon D, Gleed RD, Dobson A. Accuracy of dilution techniques for access flow measurement during hemodialysis. Am J Kidney Dis. 1998 Mar;31(3):502-8. doi: 10.1053/ajkd.1998.v31.pm9506688.
- [Background] Vesely TM, Gherardini D, Gleed RD, Kislukhin V, Krivitski NM. Use of a catheter-based system to measure blood flow in hemodialysis grafts during angioplasty procedures. J Vasc Interv Radiol. 2002 Apr;13(4):371-8. doi: 10.1016/s1051-0443(07)61739-4. PMID 11932367